CLINICAL TRIAL: NCT06961513
Title: Patient-reported Outcomes and Views of Treatments for Pelvic-floor Muscle Dysfunction, and Their Relationship to Patient Psycho-social Characteristics.
Brief Title: Patient Evaluation of Treatment of Pelvic-floor Muscle Dysfunction.
Status: Not yet recruiting | Type: Observational
Sponsor: Swansea University (Other)
Responsible Party: Sponsor
Other Study IDs: 12645
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Pelvic-floor Disorders
Keywords: Pelvic-floor disorders; patient views; Women's health physiotherapy; psychology
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with pelvic-floor muscle dysfunction: Women with pelvic-floor muscle dysfunction undergoing women's health physiotherapy
  Interventions: Other: Women's health physiotherapy

INTERVENTIONS:
Other: Women's health physiotherapy — Women's health physiotherapy for pelvic-floor dysfunction

SUMMARY:
Pelvic-floor muscle dysfunction (PFMD) affects 25% of women. It involves urinary and faecal incontinence, prolapse, sexual dysfunction, pelvic pain, and is associated with psycho-social issues (depression, anxiety), impacting negatively quality-of-life. First-line treatment for PFMD is women's health physiotherapy, which is safe, patient acceptable, and clinically effective. However, its effectiveness can be compromised by patient nonattendance/nonengagement, which can result in worsening of condition necessitating later surgery. The current research assesses factors contributing to outcomes, and nonattendance/nonengagement, so this knowledge may help improve healthcare system support and delivery. A range of routinely-collected factors at intake (physical functioning, psychological functioning, and demographic-social characteristics) will be related to routinely-gathered outcomes (patient-rated improvement in function; attendance and engagement). Additionally, a subset of patients who either attended or did not attend appointments, will be interviewed about their reasons for attendance/nonattendance. The aims are to determine: (1) whether any patient factors predict outcomes (functioning, attendance/engagement); (2) whether clusters of intake-factors differentiate patients who did/did not attended; and (3) patient views on why they attended or did not. Consecutively referred women with PFMD at the Women's Health Unit, Singleton Hospital, Swansea, will be asked for informed consent to participate. Following consent, routine assessment height, weight, age, diagnosis any physical measures of pelvic floor functioning will be taken, collected by medical staff. Questionnaires on patient-reported measures of pelvic-function, general health, quality of life, and psychological state will be completed, which should take 30min to complete. Patients will then have physiotherapy treatment, as usual. At discharge, the same data will be obtained. A subset of patients (N=80) will be contacted following initial appointment; half who attended, and half who did not. Following their consent to a telephone interview concerning their thoughts on the healthcare offered, and reasons they did/did not attend. This interview will be conducted, recorded anonymously, and analysed.

DETAILED DESCRIPTION:
Approximately 700 women with pelvic-floor muscle dysfunction (PFMD), consecutively referred to the Women's Health Unit at Singleton Hospital, Swansea, will be given full information about the study at their initial referral at Singleton Hospital, and asked if they would consent to participate. Following consent, routine assessment height, weight, age, diagnosis any physical measures of pelvic floor functioning will be taken, collected by medical staff The participants will ask completed questionnaires around patient-reported measures of their pelvic-function (Queensland), general health (SF-12) quality of life (EQ-5D), and psychological state (HADS; PVQ-II; ACEs; LSI; WPAQ) questionnaires. The should take about 30 minutes to complete. Patients will then have their Women's Health Physiotherapy treatment, as usual, which will not be impacted this research. At discharge, the same data as described above will be obtained. A randomly selected subset of patients (N=80) will be contacted following their initial appointment. Half of these will have attended, and half will not have attended their interview. Following them giving their informed consent to a telephone interview, they will participate in a semi-structured interview concerning their thoughts on the healthcare offered, and reasons they did/did not attend. This interview will last 15-30 minutes, depending on the participant, be conducted by a researcher who is not a member of their healthcare team, recorded anonymously, and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Over 18 years old
* Diagnosed with pelvic floor muscle dysfunction
* Patients referred for physiotherapy treatment at the Women's Health Unit of Singleton Hospital, Swansea

Exclusion Criteria:

* Patients under 18
* Patients who don't have PFMD
* Patients unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 years of age with pelvic-floor disorders
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-04-29 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Attendance at sessions and improvement in pelvic-floor function. | 5 years
  Attendance at scheduled sessions will be recorded, as will change in routinely collected pelvic floor functioning data.

CONTACTS AND LOCATIONS:
Locations (1):
- Singleton Hospital, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No sharing will be needed outside the research team.